CLINICAL TRIAL: NCT03955731
Title: Optical Coherence Guided Treatment of ST-segment Elevation Myocardial Infarction With the Drug-eluting Resorbable Magnesium Scaffold: the BEST- MAG Multicentre Study. (BElgian ST-segment Elevation Myocardial Infarction Treatment With Resorbable MAGnesium Scaffold).
Brief Title: OCT Guided Magmaris RMS in STEMI
Acronym: BESTMAG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Centre Hospitalier Universitaire Saint Pierre (Other); Universitair Ziekenhuis Brussel (Other); CHU de Charleroi (Other); Jolimont (Unknown); Ziekenhuis Oost-Limburg (Other); University Hospital St Luc, Brussels (Other); Centre Hospitalier Universitaire UCLouvain Namur (Other); Le centre hospitalier EpiCURA (Unknown); Centre Hospitalier Régional de la Citadelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 62036
Record Dates: First submitted 2019-02-11; First posted 2019-05-20 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single study arm (Other): STEMI Patients treated with Magmaris resorbable magnesium scaffold
  Interventions: Device: Magmaris resorbable magnesium scaffold

INTERVENTIONS:
Device: Magmaris resorbable magnesium scaffold — Implantation of Magmaris resorbable magnesium scaffold

SUMMARY:
Percutaneous treatment of coronary artery disease depends on the implantation of stents within diseased coronary segments. Compared with conventional bare-metal and drug- eluting stents, which remain permanently within the coronary anatomy, bioresorbable scaffolds (BRS) offer several potential advantages due to its resorbable properties. The resorbable magnesium scaffold Magmaris has demonstrated favourable outcomes in patients with stable coronary artery disease. In particular, in comparison to polymeric bioresorbable scaffolds, no cases of stent thrombosis have been reported in over two years of follow-up suggesting that magnesium-based resorbable scaffolds have low thrombogenicity and might be particularly beneficial for patients presenting with ST- segment myocardial infarction. A recent pilot study in eighteen patients supports this concept, which has led to the development of the proposed prospective multicentre study including intra-coronary imaging with long-term clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with a ST-elevation myocardial infarction (STEMI) with symptoms onset <24 hours or with ongoing symptoms.
2. Signed patient informed consent.

Exclusion Criteria:

1. Age < 18 or > 70 years.
2. Pregnancy or breastfeeding.
3. Cardiogenic shock.
4. Creatinine clearance ≤30 ml/min/1.73 m2 (as calculated by MDRD formula for estimated GFR) and not on dialysis. Note: chronic dialysis dependent patients are eligible for enrolment regardless of creatinine clearance.
5. Infarct-artery reference diameter < 2.7 or > 4.0 mm (within the segment of the culprit lesion) by visual estimation, and OCT infarct-artery distal reference mean lumen diameter < 2.7 or > 3.7 mm
6. Non-optimal vessel preparation after predilatation: residual stenosis >30%.
7. Culprit lesion length > 21 mm.
8. Culprit lesion located within a previously stented segment (stent thrombosis or in-stent restenosis).
9. Culprit lesion involving a saphenous vein graft.
10. Culprit lesion involving a bifurcation with an intended two-stent implantation strategy.
11. Ostial right coronary artery
12. Severe calcification or tortuosity of the infarct-related artery.
13. Absolute contraindication to a 12 months dual antiplatelet therapy.
14. Life expectancy < 3 years.
15. Patients taking oral anticoagulant therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-02-15 (Actual); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
A device oriented composite endpoint (DOCE) including cardiac death, target vessel myocardial infarction (attributable to the culprit lesion) and ischemic-driven target lesion revascularization (TLR) within 12 months after the index procedure. | 1 year
  DOCE at 12 months

SECONDARY OUTCOMES:
Procedural success defined as the delivery and deployment of RMS at the intended target lesion with a final residual stenosis ≤20% by visual estimation. | in-hospital
  Procedure succes
DOCE at 1-,6- and 24-months follow-up periods. | 2 years
  DOCE at 1,6 and 24 months
Definite or probable scaffold thrombosis. | 2 years
  incidence scaffold thrombosis
Vessel healing assessment through an angiographic with OCT follow- up procedure at 15 months in predetermined participating centres | 15 months
  Healing characteristics on OCT evaluation
All-cause death, cardiac death, non-TVR, any revascularization at 1, 6, 12 and 24 months. | 2 years
  MACE

CONTACTS AND LOCATIONS:
Locations (1):
- Johan Bennett, Leuven, Brabant, Belgium